CLINICAL TRIAL: NCT03661268
Title: The Effect of Rapid Fluid Challenge Under Pulmonary Artery Catheter Monitoring on Physiological Indexes of Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Fifth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002(yan)-02
Record Dates: First submitted 2018-09-02; First posted 2018-09-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: A bag of 500ml of normal saline is infused within 15 minutes using a bag pressurized to 300 mmHg. All other treatments, including maintenance fluids, dose of vasoactive agents and ventilator settings, remain unchanged during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Septic shock (Experimental): Patients (at least 18 years of age, no more than 75 years old) with refractory hypotension secondary to sepsis who, at the discretion of treating physicians, required fluid challenge in the presence of pulmonary artery catheter. Refractory hypotension was defined as need of vasopressors to maintain systolic blood pressure (SBP) no less than 90 mmHg despite adequate fluid resuscitation.
  Interventions: Other: fluid chanllenge

INTERVENTIONS:
Other: fluid chanllenge — A bag of 500ml of normal saline is infused within 15 minutes using a bag pressurized to 300 mmHg.

SUMMARY:
Fluid challenge is often carried out in septic shock patients. Its responsiveness usually requires invasive monitoring. The pulmonary artery catheter(PAC) is the most effective means of monitoring.To use non-invasive methods is very tempting. Investigators hypothesize that venous-to-arterial carbon dioxide difference,venous-to-arterial carbon oxygen difference, central venous-arterial carbon dioxide to arterial-venous oxygen content ratio and Central Venous SO2 variations provides feasible estimation on fluid responsiveness in septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old; less than 75 years old ICU patients
* Septic shock
* Monitored with pulmonary artery catheter (Swan-Ganz catheter)
* The decision of fluid challenge made by the treating physician

Exclusion Criteria:

* Evidence of fluid overload
* Pregnancy
* Recently participated in other studies
* Severe heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
cardiac index change | Immediately after fluid challenge
  Fluid responsiveness: increase in CI of at least 10% after fluid challenge ;Fluid nonresponsiveness:no increase or increase in CI less than 10%.

CONTACTS AND LOCATIONS:
Overall Officials: wang ping, MD, Study Chair — Chengdu Fifth People's Hospital
Locations (1):
- ICU of Chengdu Fifth People's Hospital, Chengdu, Sichuan, China